CLINICAL TRIAL: NCT01158716
Title: Remote Ischemic Preconditioning in ad Hoc Percutaneous Coronary Interventions: a Randomized Clinical Study
Brief Title: Remote Ischemic Preconditioning in ad Hoc Percutaneous Coronary Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiovascular Research Society, Greece (Other)
Responsible Party: Principal Investigator, Dr D Katritsis, Head of Department of Cardiology, Athens Euroclinic, Cardiovascular Research Society, Greece
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4.7.7.2010
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Results first posted 2014-04-09 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-03

CONDITIONS: Coronary Artery Disease
Keywords: percutaneous coronary intervention; remote ischemic preconditioning
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote Ischemic Preconditioning (Active Comparator)
  Interventions: Other: Remote Ischemic Preconditioning
- Control (No Intervention)

INTERVENTIONS:
Other: Remote Ischemic Preconditioning — Patients are subjected to a 5-minute ischemia of the non-dominant arm with the use of a blood pressure cuff (inflated at 200mm Hg)
  Arms: Remote Ischemic Preconditioning

SUMMARY:
Elective percutaneous coronary intervention (PCI) is associated with troponin release in approximately one third of cases. Myocardial necrosis may result from downstream embolization of atheromatous material, coronary side-branch occlusion and may involve ischemia/reperfusion injury. The investigators hypothesized that a single remote ischemic preconditioning cycle would reduce peri-procedural troponin release.

DETAILED DESCRIPTION:
Elective percutaneous coronary intervention (PCI) is associated with troponin release in approximately one third of cases, which is a sensitive and specific marker of myocyte necrosis. Myocardial necrosis may result from downstream embolization of atheromatous material, coronary side-branch occlusion and may involve ischemia/reperfusion injury. A number of studies have demonstrated that procedure-related troponin release is associated with subsequent cardiovascular events and a worst prognosis, especially in those patients with the most marked elevation in troponin concentration.

Recently, 3 cycles of 5-minute ischemia followed by 5-minute reperfusion of the upper extremities were shown to reduce troponin release in elective PCI. However, this ischemic preconditioning (IPC) protocol requires 30 minutes and is of limited use in the context of PCI at the time of initial cardiac catheterization (ad hoc coronary intervention).

Since experimental evidence suggests that IPC is a graded than an "all-or-nothing" phenomenon, and even a short, single IPC cycle may have protective effects in the myocardium, the investigators hypothesized that patients undergoing ad hoc coronary intervention would have reduced peri-procedural troponin release if subjected to a single, remote IPC cycle, between diagnostic catheterization and coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a significant stenosis as documented in coronary angiography eligible for PCI
* Patients ≥ 18 of age and able to give informed consent

Exclusion Criteria:

* Severe comorbidity (estimated life expectancy <6 months)
* Use of nicorandil or glibenclamide
* Elevated baseline cTnI before PCI
* Renal disease as documented by serum creatinine before PCI
* LVEF<35%

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Demosthenes G Katritsis, MD, PhD, Study Chair — Athens Euroclinic
Locations (1):
- Athens Euroclinic, Athens, Attica, Greece

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Remote Ischemic Preconditioning | Control
Started | 48 | 48
Completed | 47 | 47
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remote Ischemic Preconditioning | Control | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (10.4) | 60.2 (10.9) | 60.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 42 | 41 | 83

OUTCOME MEASURES:

1. Primary Outcome: Delta Cardiac Troponin I (ΔcTnI)
Description: ΔcTnI is defined as cardiac troponin I (cTnI) at 24 hours post-PCI minus cTnI before coronary angiography
Time Frame: 24 hours post PCI
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Remote Ischemic Preconditioning | Control
Number analyzed (Participants) | 47 | 47
ng/mL | 0.04 [0.01 to 0.14] | 0.19 [0.18 to 0.59]

2. Secondary Outcome: Chest Pain During Coronary Balloon Occlusion
Description: Chest pain severity was assessed with a 10 point scale (0: no pain, 10: most severe discomfort ever experienced)
Time Frame: During coronary balloon occlusion
Reporting Status: Not Posted

3. Secondary Outcome: ECG Evidence of Ischemia During Coronary Balloon Occlusion
Description: ST-segment deviation as monitored during coronary balloon occlusion
Time Frame: During coronary balloon occlusion
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Remote Ischemic Preconditioning | Control
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 0/47 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No